CLINICAL TRIAL: NCT02176382
Title: Denosumab and Teriparatide Study (DATA-HD and DATA-EX)
Acronym: DATA-HD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Benjamin Leder, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014P000853
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Denosumab; Teriparatide; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard dose teriparatide (Active Comparator): teriparatide daily subcutaneous injection (months 0-9) plus denosumab subcutaneous injection every 6 months (months 3-15) followed by zoledronic acid at month 15
  Interventions: Drug: denosumab; Drug: teriparatide; Drug: Zoledronic acid
- High dose teriparatide (Active Comparator): teriparatide alternate dose daily subcutaneous injection (months 0-9) plus denosumab subcutaneous injection every 6 months (months 3-15) followed by zoledronic acid at month 15
  Interventions: Drug: denosumab; Drug: teriparatide; Drug: Zoledronic acid

INTERVENTIONS:
Drug: denosumab — denosumab subcutaneous injection
  Other Names: Prolia
Drug: teriparatide — teriparatide daily subcutaneous injection
  Other Names: Forteo
Drug: Zoledronic acid — zoledronic acid infusion
  Other Names: Reclast

SUMMARY:
The aim of the study is to assess the effect of an antiresorptive medication in combination with standard dose or alternate dose teriparatide. The study extension will evaluate the effect of one-dose of zoledronic acid after the teriparatide/denosumab combination.

ELIGIBILITY:
Inclusion Criteria:

* women aged 45+
* postmenopausal
* osteoporotic with high risk of fracture

Exclusion Criteria:

* no significant previous use of bone health modifying treatments

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-08; Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Leder, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Ramchand SK, David NL, Leder BZ, Tsai JN. Bone Mineral Density Response With Denosumab in Combination With Standard or High-Dose Teriparatide: The DATA-HD RCT. J Clin Endocrinol Metab. 2020 Mar 1;105(3):890-7. doi: 10.1210/clinem/dgz163. PMID 31674641
- [Background] Ramchand SK, David NL, Lee H, Bruce M, Bouxsein ML, Leder BZ, Tsai JN. Effects of Combination Denosumab and High-Dose Teriparatide Administration on Bone Microarchitecture and Estimated Strength: The DATA-HD HR-pQCT Study. J Bone Miner Res. 2021 Jan;36(1):41-51. doi: 10.1002/jbmr.4161. Epub 2020 Sep 19. PMID 32790196
- [Result] Tsai JN, Lee H, David NL, Eastell R, Leder BZ. Combination denosumab and high dose teriparatide for postmenopausal osteoporosis (DATA-HD): a randomised, controlled phase 4 trial. Lancet Diabetes Endocrinol. 2019 Oct;7(10):767-775. doi: 10.1016/S2213-8587(19)30255-4. Epub 2019 Aug 22. PMID 31447409

RESULTS

PARTICIPANT FLOW:
Period: DATA-HD Study
Arm/Group | Standard Dose Teriparatide | High Dose Teriparatide
Started | 39 | 37
Completed | 31 | 29
Not Completed | 8 | 8
Period: DATA-HD Extension
Arm/Group | Standard Dose Teriparatide | High Dose Teriparatide
Started (7 subjects completed DATA-HD but did not enroll in extension study.) | 27 | 26
Completed | 26 | 26
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Includes all subjects who completed at least 1 post-baseline visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dose Teriparatide | High Dose Teriparatide | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (7.0) | 67.0 (7.3) | 66.4 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 34 | 69
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 34 | 33 | 67
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 33 | 33 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Spine Bone Mineral Density by Dual X-ray Absorptiometry (DXA)
Time Frame: Baseline and 42 months
Population: Population includes those who completed a month 42 visit.
Measure: Mean (Standard Deviation); unit: percent change in BMD
Arm/Group | Standard Dose Teriparatide | High Dose Teriparatide
Number analyzed (Participants) | 26 | 26
percent change in BMD | 7.69 (4.66) | 12.70 (5.54)

ADVERSE EVENTS:
Time Frame: 3.5 years
Arm/Group | Standard Dose Teriparatide | High Dose Teriparatide
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/37
Serious Adverse Events (participants affected / at risk) | 9/39 | 2/37
Other Adverse Events (participants affected / at risk) | 0/39 | 2/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Dose Teriparatide (N=39) | High Dose Teriparatide (N=37)
wrist fracture (Musculoskeletal and connective tissue disorders) | 2 | 1
anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
clavicle fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
fibula avulsion fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
humeral fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
kidney cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
pancreatitis (Endocrine disorders) | 1 | 0
rib fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
shoulder dislocation (Musculoskeletal and connective tissue disorders) | 1 | 0
throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
vertebral fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Dose Teriparatide (N=39) | High Dose Teriparatide (N=37)
back pain (Musculoskeletal and connective tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT02176382/Prot_SAP_000.pdf